CLINICAL TRIAL: NCT01632631
Title: Patient-specific Virtual Reality Rehearsal Prior to EVAR: Influence on Technical and Non-technical Operative Performance. A Randomized Controlled Trial.
Brief Title: Patient-specific Virtual Reality Rehearsal Prior to EVAR: Influence on Technical and Non-technical Operative Performance
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2012/412
Record Dates: First submitted 2012-06-28; First posted 2012-07-03 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Infrarenal Aortic Aneurysm
Keywords: suitable for endovascular exclusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PROcedure rehearsal: PROcedure rehearsal performed before real EVAR procedure No intervention
- No PROcedure rehearsal: no PROcedure rehearsal performed before real EVAR procedure No intervention

SUMMARY:
Ongoing technological advances, especially in the field of image processing, have refined medical simulations to offer life-like replications of medical and surgical procedures in a variety of specialties. Patient-specific image data are incorporated into these simulations, and transformed into a 3D model. This enables the practitioner and his/her team to perform and practice 'real' cases on a virtual patient prior to performing the real procedure on the actual patient. This new technology has been referred to as 'patient-specific' rehearsal, also 'mission' or 'procedure' rehearsal.

Research has already proven that simulated patient-specific rehearsal of a carotid artery stenting procedure may enhance surgical and team performance.

The PROcedure rehearsal software can now also be used to practice patient-specific endovascular repair of infrarenal aortic aneurysms (EVAR). The ability to rehearse a challenging and complex procedure like EVAR may not only influence device selection based on preoperative planning, but also improve the technical performance of the surgeon/radiologist and the awareness and communication within the entire endovascular team. However, further research is needed to evaluate if this new technology may enhance clinical safety and efficiency, i.e. if patients actually benefit from physicians and team members conducting patient-specific rehearsals of EVAR interventions.

ELIGIBILITY:
Inclusion Criteria:

-infrarenal aortic aneurysm suitable for endovascular exclusion

Exclusion Criteria:

* Adult patients who do not have capacity to consent.
* Previous stent-graft implanted in the abdominal aorta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an infrarenal aortic aneurysm suitable for endovascular exclusion. The suitability for endovascular repair is based upon the physician's decision.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Technical operative metrics | during EVAR procedure
  * C-arm positioning for proximal and distal landing zone
  * Fluoroscopy time
  * Number of angiograms
  * Amount of contrast
Errors occurring during EVAR procedure (Imperial College Error Capture record) | during EVAR procedure

SECONDARY OUTCOMES:
Subjective sense of realism of patient-specific rehearsal reported by team members | immediately after EVAR procedure
  Subjective sense of realism of patient-specific rehearsal reported by team members (Measurement: questionnaire)
Team satisfaction | immediately after EVAR procedure
  Team satisfaction Measurement: questionnaire
Any deviation from initial treatment plan | immediately after EVAR procedure
30 day mortality and morbidity | within the first 30 days after surgery
Technical and clinical success rate | immediately after EVAR procedure
  * Successful access to the arterial system using a remote site
  * Successful deployment of the endoluminal graft with secure proximal and distal fixation
  * Absence of either type I or III endoleak
  * Patent endoluminal graft without significant twist, kinks, or obstruction
Initial clinical success | within the first 30 days after surgery
  o Successful deployment of the endovascular device at the intended location, without:
  * Death as a result of aneurysm-related treatment
  * Type I or III endoleak
  * Graft infection or thrombosis
  * Aneurysm expansion (diameter > 5mm)
  * Aneurysm rupture
  * Conversion to open repair
  * Graft dilatation (≥ 20% by diameter)
  * Graft migration
  * Failure of device integrity

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Desender, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (2):
  - Sint - Maarten Hospital, Campus Rooienberg, Duffel
  - Ghent University Hospital, Ghent
- Zurich University Hospital, Zurich, Switzerland

REFERENCES:
- [Derived] Desender L, Van Herzeele I, Lachat M, Duchateau J, Bicknell C, Teijink J, Heyligers J, Vermassen F; PAVLOV Study Group. A Multicentre Trial of Patient specific Rehearsal Prior to EVAR: Impact on Procedural Planning and Team Performance. Eur J Vasc Endovasc Surg. 2017 Mar;53(3):354-361. doi: 10.1016/j.ejvs.2016.12.018. Epub 2017 Jan 20. PMID 28117241